CLINICAL TRIAL: NCT01506765
Title: Schizophrenia, Related Troubles and Glutathione: Clinical Trial. Effects of Oral Administration of N-Acetylcysteine (NAC) on the Brain Glutathione Level and on the Symptoms of Schizophrenia: Double-blind and Crossover Study
Brief Title: Schizophrenia, Related Troubles and Glutathione: Clinical Trial. Effects of Oral Administration of N-Acetylcysteine (NAC) on the Brain Glutathione Level and on the Symptoms of Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Dresse Kim Q. Do, Professor, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 106/03 CE
Record Dates: First submitted 2012-01-03; First posted 2012-01-10 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2012-01

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; glutathione; NAC; Neurological scales; Magnetic Resonance Spectroscopy (MRS); EEG/evoked potentials; fibroblasts; patients who receive NAC; patients who receive placebo
MeSH Terms: conditions — Schizophrenia | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- patients who receive NAC first (Active Comparator): this group will receive 2g/day of NAC (2 caps of 0.5g twice day)for a duration of 8 weeks first, and after this 8 weeks their receive placebo for 8 weeks.
  Interventions: Drug: N-Acetyl-Cysteine (NAC)
- patients who receive placebo first (Placebo Comparator): this patients will receive first placebo for a duration of 8 weeks, and after this 8 weeks their receive NAC for 8 weeks
  Interventions: Drug: N-Acetyl-Cysteine (NAC)

INTERVENTIONS:
Drug: N-Acetyl-Cysteine (NAC) — Once included, the patients will be randomly placed in two groups: one group (1) will receive 2 g/day of NAC (2caps of 0.5g twice a day) and the other group (2) a placebo, for a duration of 8 weeks. At the end of the 8 weeks, group (2) will receive NAC and (1) the placebo for another 8 weeks

SUMMARY:
The results of the study "schizophrenia, related disorders and glutathione" conducted at the Laboratory of Psychiatric Neuroscience (LUNEP) DUPA of Lausanne, reinforce the hypothesis proposed that a deficit intracerebral glutathione is a vulnerability factor for Schizophrenia at least for a subgroup of patients. While pursuing the baseline study, it is appropriate now to try to restore a higher level of glutathione in patients to see if this increase is accompanied by an improvement in symptoms, particularly negative symptoms and disorders cognitive, particularly resistant to current therapy. N-acetyl-cystein (NAC) is a precursor of glutathione which is used clinically for various indications, well tolerated even at high doses. The investigators propose a double-blind cross-over with the aim to study if the N-acetyl-cystein (at a dose of oral 2g/day) leads on the one hand a rising glutathione brain (measured in resonance magnetic spectroscopic) and also improved patients' conditions (determined by clinical assessments, psychopathological, neuropsychological, biochemical and physiological), while recording any side effects. As a first step, this study should include at least thirty patients and last for two to three years. It is important to note that this is not a study of medication suggested by a pharmaceutical industry, but a medical search.

DETAILED DESCRIPTION:
The results of the study "schizophrenia, related disorders and glutathione" conducted at the Laboratory of Psychiatric Neuroscience (LUNEP) DUPA of Lausanne, reinforce the hypothesis proposed that a deficit intracerebral glutathione is a vulnerability factor for Schizophrenia at least for a subgroup of patients. While pursuing the baseline study, it is appropriate now to try to restore a higher level of glutathione in patients to see if this increase is accompanied by an improvement in symptoms, particularly negative symptoms and disorders cognitive, particularly resistant to current therapy. N-acetyl-cysteine (NAC) is a precursor of glutathione which is used clinically for various indications, well tolerated even at high doses. The investigators propose a double-blind cross-over with the aim to study if the N-acetyl-cystein (at a dose of oral 2g/day) leads on the one hand a rising glutathione brain (measured in resonance magnetic spectroscopic) and also improved patients' conditions (determined by clinical assessments, psychopathological, neuropsychological, biochemical and physiological), while recording any side effects. As a first step, this study should include at least thirty patients and last for two to three years. It is important to note that this is not a study of medication suggested by a pharmaceutical industry, but a medical search.

ELIGIBILITY:
Inclusion Criteria:

* patients (male or female, aged 18 to 65 years, QI>70) meeting the DSM-IV criteria (established by a senior psychiatrist) for schizophrenia and have the capacity to consent to the study. The study population include both inpatients and outpatients who are currently taking at least one of the following:Olanzapine, Clozapine, Haloperidol, Risperidone, Flupenthixol, or Fluphenazine. The following guidelines have been established for potential medication changes that patients may undergo during the course of the trial.
* dose changes to existing medication (either increases or decreases in dose) will be accepted and participants will be allowed to continue with the trial.
* A change in primary antipsychotics from one medication to another will require participants to withdrawn from the study.
* An addiction of another antipsychotic, secondary to the existing antipsychotic treatment (primary antipsychotic) will be acceptable providing that there isn't a complete change from one antipsychotic to another.

Exclusion Criteria:

* pregnancy
* acute psychotic state, preventing the patient cooperation
* co-morbidity with drug dependency
* organic cerebral disease, major somatic diseases
* abnormal renal, hepatic, thyroid or hematological findings
* treatment with a regulator of mood(lithium, valproate, topiramate, lamotrigine et carbamazepine)
* allergy to NAC
* treatment with antioxidants

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2003-08; Primary Completion 2004-12 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Positive and Negative Syndrome Scale (PANSS) | 8 months
  Improvment of the negative symptoms, measured with the PANSS: positive and negative syndrome scale". (Score:1= absence of the symptom - 7= extreme symptoms)

SECONDARY OUTCOMES:
frankfurt Complaint Questionnaire (FCQ) | 8 months
  Assessment of subjective troubles, " basic symptoms ": troubles of perceptive, cognitive or motor functions frequently observed in prodromal or remission phases.
Global Assessment of Functioning - (GAF) | 8 months
  Assessment of the psychological, social and professional state of the patient at a given moment.
Clinical Global Impression - (CGI) | 8 months
  Allows punctual evaluation of the severity of the disease, of the improvement and of the side effects
Neuropsychological evaluation | 8 months
  The neuropsychological tests aim to assess cognitive functions : working memory, attention, planning; also include a WAIS
Neurological scales for the assessment of extrapyramidal symptoms | 8 months
  AIMS (Abnormal Involuntary Movements Scale): quantitative assessment of secondary hyperkinesia (excluding tremor) due to neuroleptics.
• Magnetic Resonance Spectroscopy (MRS) | 8 months
  A MRS method has originally been developed for the determination of brain GSH levels in vivo (Trabesinger et al., 1999), allowing us to observe a 51% GSH decrease in prefrontal cortex of schizophrenic patients (Do et al., 2000).
EEG/evoked potentials | 8 months
  Anomalies of amplitude and latency of the P300 wave evoked under the "auditory oddball" paradigm are reliable neurophysiological markers of schizophrenia, correlating with the negative symptoms
Blood and fibroblasts biochemistry | 8 months
  I. Plasma GSH and metabolites, plasma amino acids, particularly the sulfur containing ones II. activity of enzymes involved in GSH metabolism III. genetic analysis of enzymes involved in GSH metabolism IV. cell counts and tests of hepatic, renal and thyroid functions
Neurological scales for the assessment of extrapyramidal symptoms | 8 months
  Simpson-Angus scale for extrapyramidal signs: tremor, rigidity, akinesia.
Neurological scales for the assessment of extrapyramidal symptoms | 8 months
  Barnes scale: specific assessment of akathisia.

CONTACTS AND LOCATIONS:
Overall Officials: Kim Do, Professor, Study Director — CNP/ LUNEP

REFERENCES:
- [Background] Do KQ, Trabesinger AH, Kirsten-Kruger M, Lauer CJ, Dydak U, Hell D, Holsboer F, Boesiger P, Cuenod M. Schizophrenia: glutathione deficit in cerebrospinal fluid and prefrontal cortex in vivo. Eur J Neurosci. 2000 Oct;12(10):3721-8. doi: 10.1046/j.1460-9568.2000.00229.x. PMID 11029642
- [Background] Mathalon DH, Ford JM, Pfefferbaum A. Trait and state aspects of P300 amplitude reduction in schizophrenia: a retrospective longitudinal study. Biol Psychiatry. 2000 Mar 1;47(5):434-49. doi: 10.1016/s0006-3223(99)00277-2. PMID 10704955
- [Background] Terpstra M, Henry PG, Gruetter R. Measurement of reduced glutathione (GSH) in human brain using LCModel analysis of difference-edited spectra. Magn Reson Med. 2003 Jul;50(1):19-23. doi: 10.1002/mrm.10499. PMID 12815674
- [Background] Trabesinger AH, Weber OM, Duc CO, Boesiger P. Detection of glutathione in the human brain in vivo by means of double quantum coherence filtering. Magn Reson Med. 1999 Aug;42(2):283-9. doi: 10.1002/(sici)1522-2594(199908)42:23.0.co;2-q. PMID 10440953
- [Derived] Carmeli C, Knyazeva MG, Cuenod M, Do KQ. Glutathione precursor N-acetyl-cysteine modulates EEG synchronization in schizophrenia patients: a double-blind, randomized, placebo-controlled trial. PLoS One. 2012;7(2):e29341. doi: 10.1371/journal.pone.0029341. Epub 2012 Feb 22. PMID 22383949